CLINICAL TRIAL: NCT00859313
Title: An Open-Label Functionality, Safety, and Efficacy Study of the NanoTab® Delivery System/ARX-F01 15 Mcg in Patients Undergoing Elective Unilateral Knee Replacement
Brief Title: An Open-Label Functionality, Safety and Efficacy Study in Patients Undergoing Elective Unilateral Knee Replacement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Talphera, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARX-C-004
Record Dates: First submitted 2009-03-09; First posted 2009-03-11 (Estimated); Results first posted 2012-02-27 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sufentanil NanoTab PCA System/15 mcg (Experimental)
  Interventions: Drug: Sufentanil NanoTab PCA System/15 mcg

INTERVENTIONS:
Drug: Sufentanil NanoTab PCA System/15 mcg — 15 mcg Sufentanil NanoTab taken sublingually q 20 minutes as needed for pain for 12 hours

SUMMARY:
This study is being performed to evaluate the functionality of a device (Sufentanil NanoTab® PCA System) that has been developed for use by patients to self-administer the ARX-F01 pain medication (Sufentanil NanoTab 15 mcg) for the treatment of post-operative pain after undergoing knee replacement surgery.

Another goal of this study is to assess the safety and effectiveness of this non-invasive, sublingual route of administration of ARX-F01 in decreasing the amount of pain that a patient experiences following knee replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between 45 and 80 years of age.
2. Patient is scheduled for an elective unilateral, unicondylar, bi- or tri-compartmental, cemented or uncemented knee replacement under general or spinal anesthesia that does not include use of an intrathecal opioid.
3. Patient must be classified as American Society of Anesthesiologists (ASA) class I - III.
4. Patient must have a Body Mass Index (BMI) between 18 and 39, inclusively.
5. Female patients of childbearing potential must be using an effective method of birth control from the screening visit through the end of study. Acceptable methods of birth control include oral or transdermal contraceptives, condom, spermicidal foam, intrauterine device (IUD), progestin implant or injection, abstinence, vaginal ring, or sterilization of partner. The reason for non-childbearing potential, such as bilateral tubal ligation, bilateral oophorectomy, hysterectomy, or postmenopausal for ≥1 year, must be specified in the patient's CRF.
6. The patient must be willing and able to understand the study procedures and the use of pain scales, and to communicate meaningfully with the study personnel.
7. The patient must have the manual dexterity to handle the Sufentnail NanoTab PCA System and be able to follow directions for its use.
8. The patient must provide written informed consent and sign the Informed Consent approved by the Institutional Review Board (IRB).

Exclusion Criteria:

1. Patient has previously undergone a knee replacement of the same knee.
2. A passive range-of-motion (PRM) will be used before the 12-hour study period is complete.
3. Patient has previously not responded to opioid analgesics for treatment of pain.
4. Patient is currently taking or has taken an opioid for more than 30 consecutive days of daily use at a daily dose equivalent of greater than 15 mg morphine within the past three months prior to surgery (e.g. more than 3 doses per day of Vicodin®, Norco®, Lortab® with 5 mg hydrocodone per tablet).
5. Patient has an allergy or hypersensitivity to opioids.
6. Patient is taking monoamine oxidase inhibitors (MAOIs), or has taken MAOIs within 14 days prior to enrolling in the study.
7. Patient currently has sleep apnea that has been documented by a sleep laboratory study.
8. Patient has any screening laboratory test value outside the laboratory normal range which is considered clinically significant by the Investigator.
9. Patient is a woman who is pregnant or lactating.
10. Patient has psychiatric disease or encephalopathy severe enough to prevent patient from providing reliable study documentation.
11. Patient, in the Investigator's judgment, does not have adequate ability to read and understand English.
12. Patient has a medical condition that, in the Investigator's opinion, could adversely impact the patient's participation or safety, conduct of the study, or interfere with the pain assessments, including fracture or active infection.
13. Patient has clinically significant renal or liver impairment which could affect metabolism or clearance of sufentanil.
14. Patient has a painful physical condition other than knee arthritis that, in the opinion of the Investigator, may confound post-operative pain assessments.
15. Patient has a history of drug, prescription medicine, or alcohol abuse within the past 2 years or a positive drug screen test for cocaine, amphetamines, barbiturates, phencyclidine, or methadone at screening.
16. Patient is receiving oxygen therapy at the time of screening.
17. Patient participated in a clinical trial of an investigational drug or device within 30 days of screening visit or is scheduled to receive an investigational product other than the Sufentanil NanoTab PCA System while participating in this study.

Exclusion Criteria Prior to Treatment Initiation:

1. Patient has a respiratory rate that is less than 8 breaths per minute or greater than 24 breaths per minute.
2. Patient has arterial oxygen saturation by pulse oximetry (SpO2) of less than 90% with supplemental oxygen.
3. Patient is not able to answer questions and follow commands.
4. Patient has vomiting that is not responsive to standard treatment.
5. The surgical procedure from incision to closure lasted more than 3 hours.
6. There have been any deviations from the surgical or anesthetic protocols as specified in Section 6.1.2.1.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela P Palmer, MD PhD, Study Director — Talphera, Inc
Locations (3):
- United States (3):
  - West Alabama Research, Inc, Birmingham, Alabama
  - Orthopedic Center of Vero Beach, Vero Beach, Florida
  - Memorial Hermann/Memorial City Medical Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Sufentanil NanoTab PCA System/15 Mcg: 15 mcg Sufentanil NanoTab taken sublingually q 20 minutes as needed for 12 hours
Period: Overall Study
Arm/Group | Sufentanil NanoTab PCA System/15 Mcg
Started | 30
Completed | 26
Not Completed | 4
Not completed — Lack of Efficacy | 2
Not completed — Adverse Event | 1
Not completed — staff error | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sufentanil NanoTab PCA System/15 Mcg
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 19
Age Continuous [Mean (Standard Deviation); unit: years] | 65.7 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Without Device Failure
Description: Percent of patients who completed the study without a device failure. A device failure is defined as the failure to dispense a NanoTab, dispensing more than one NanoTab, or dispensing a broken NanoTab. Device failures were monitored and reported by study staff.
Time Frame: 12 hours
Measure: Number; unit: percent
Arm/Group | Sufentanil NanoTab PCA System/15 Mcg
Number analyzed (Participants) | 30
percent | 100

ADVERSE EVENTS:
Arm/Group | Sufentanil NanoTab PCA System/15 Mcg
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 9/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sufentanil NanoTab PCA System/15 Mcg (N=30)
nausea (Gastrointestinal disorders) | 5 (5) — possibly or probably related
vomiting (Gastrointestinal disorders) | 6 (6) — possibly or probably related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
no publication without prior written consent